CLINICAL TRIAL: NCT03350802
Title: Usefulness of Procalcitonin Test to Differentiate the Cause of Pneumonia in Patients With Cancers
Brief Title: Procalcitonin Test for Differentiation of the Cause of Pneumonia
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Hee Seok Lee, Pulmonologist, National Cancer Center, Korea
Other Study IDs: NCC2014-0018
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Procalcitonin; Pneumonia; Cancer
MeSH Terms: conditions — Pneumonia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- procalcitonin pneumonia cohort: Patients who are suspected of acute pneumonia due to symptoms and imaging findings compatible with pneumonia can be enrolled in this cohort.
  Interventions: Diagnostic Test: procalcitonin test

INTERVENTIONS:
Diagnostic Test: procalcitonin test — All patients enrolled in this cohort undergo procalcitonin test in addition to basic microbiological test.

SUMMARY:
The purpose of this study is to evaluate the usefulness of procalcitonin test for differentiation of the cause of pneumonia in patients with cancer.

DETAILED DESCRIPTION:
Serum procalcitonin test is currently used as the biomarker for bacterial infection. Especially, procalcitonin test has been reported to be helpful in differentiating bacterial pneumonia from viral pneumonia, acute exacerbations of interstitial pneumonitis or chronic obstructive lung disease. However, it is not known whether procalcitonin test can help distinguish bacterial pneumonia from non-bacterial pneumonia such as radiation pneumonitis or chemotherapy-induced pneumonitis in patients with cancer.

The aim of this prospective cohort study is to observe the clinical benefits of procalcitonin test for differentiation of the cause of pneumonia in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Patients who have symptoms and suspected imaging findings compatible with pneumonia

Exclusion Criteria:

* Patients who have been treated with antibiotics or steroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients who are suspected of acute pneumonia due to symptoms and imaging findings compatible with pneumonia can be enrolled in this cohort.
     * suspected symptom: cough, sputum, dyspnea or fever/chill
     * suspected image findings: consolidation or ground-glass opacity on chest radiograph or CT
  2. All patients enrolled in this cohort undergo procalcitonin test in addition to basic microbiological test.
     * basic microbiological test: blood culture, sputum gram stain/culture, pneumococcal urinary antigen, legionella urinary antigen, mycoplasma antibody etc.
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Procalcitonin level according to the cause of pneumonia in patients with cancer | procalcitonin level is checked within 24hours after visiting hospital
  bacterial pneumonia vs. radiation pneumonitis vs chemotherapy-induced pneumonitis

SECONDARY OUTCOMES:
Influence of neutropenia on procalcitonin level in patients with baterial pneumonia | procalcitonin level is checked within 24hours after visiting hospital
  bacterial pneumonia with neutropenia vs. without neutropenia
procalcitonin level in patients with atypical pneumonia | procalcitonin level is checked within 24hours after visiting hospital
  viral pneumonia vs tuberculosis vs fungal infection

CONTACTS AND LOCATIONS:
Overall Officials: HEE SEOK LEE, M.D., Principal Investigator — National Cancer Center
Locations (1):
- Respiratory Clinic, National Cancer Center, Goyang-si, Gyeonggi-do, South Korea